CLINICAL TRIAL: NCT02990676
Title: Exploring Computerised Cognitive Training for People With Huntington's Disease
Acronym: CogTrainHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiff University (Other)
Collaborators: Jacque and Gloria Gossweiler Foundation (Unknown); Health and Care Research Wales (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1535-16; HF-16-1152 (Other Grant/Funding Number: Health and Care Research Wales Fellowship Award to Dr. Emma Yhnell); 210821 (Other: Integrated Research Application Service Project ID)
Record Dates: First submitted 2016-09-30; First posted 2016-12-13 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Huntington's Disease
Keywords: Cognition; Computerised cognitive training; Feasibility study; Huntington's disease; Translational
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computerised cognitive training group (Experimental): Participants will be asked to complete the training programme provided using HAPPYneuron software for a minimum of 30 minutes 3 times a week for 12 weeks. The intervention will be completed in participant homes with the help of email or telephone reminders, as preferred.
  Interventions: Behavioral: Computerised cognitive training
- Control group (No Intervention): Asked to continue as normal

INTERVENTIONS:
Behavioral: Computerised cognitive training — Computerised cognitive training regime
  Arms: Computerised cognitive training group

SUMMARY:
Cognitive impairments, especially deficits of executive function, have been well documented as a core and early feature in Huntington's disease (HD). Cognitive impairments can be considerably burdensome and devastating for people and families affected by HD. Computerised cognitive training interventions that focus on improving executive function present a potentially exciting non-pharmacological treatment option. Novel work conducted in mouse models of HD, has demonstrated that cognitive training, administered from an early stage in the disease, can improve motor performance at an older age, even in the absence of further training in the intervening time. This represents proof of principle in an animal model of HD that cognitive training can improve HD disease symptoms.

Improvements associated with executive function training have also been reported in a clinical setting in a variety of neurodegenerative diseases. For example, cognitive training, can improve executive function as people age, and training specifically focused on tasks of executive function has been shown to improve both cognitive and motor outcomes in neurodegenerative diseases such as Parkinson's disease (PD) and Alzheimer's disease (AD). Therefore, this study is a feasibility study which aims to establish proof of principle for using computerised cognitive training in people with HD. The investigators propose to determine the feasibility, acceptability and gather preliminary evidence of the effectiveness of a cognitive training intervention programme, targeted for people with HD. The investigators will also aim to investigate the most appropriate outcome measures to use in this study and gather feedback on the cognitive training intervention. The investigators will also establish proof of concept via the study of brain structure and function, using MRI scanning techniques.

The computerised cognitive training software and the associated outcome measures will be investigated, taking into account the views of people and families who are affected by HD. A randomised feasibility study of computerised cognitive training for people with HD will then be conducted. Participants who are randomised to the cognitive training intervention group will be asked to complete a cognitive training intervention utilising "HAPPYneuron" software. Participants in the intervention group will be asked to complete the cognitive training programme for a minimum of 30 minutes, 3 times a week for the 12 week study duration. Participants in the control group will not receive any cognitive training and will be asked to continue as normal, however they will have home visits to control for the confounding effect of social interaction. Additional monitoring and prompting for the intervention group, will be conducted via email, text or telephone reminders (as preferred by the participant) and home visits. The motor and cognitive function of participants will be assessed at the beginning and end of the study, using a range of motor and cognitive assessments. Additional cognitive measurements will be recorded as part of the HAPPYneuron programme throughout the cognitive training intervention, such as accuracy and response time measures of particular computer games. MRI scans (optional) will be conducted at the beginning and end of the study to identify any structural changes in the brain that may be associated with the cognitive training intervention. As part of the feasibility and acceptability assessment, participants, family members and carers will be invited to complete a semi-structured interview at the end of the study, if consent is obtained, focusing on using this type of software as a home based therapeutic intervention.

DETAILED DESCRIPTION:
Due to space constraints a more extensive description of the research study can be found in the study protocol.

1. Background and Rationale Huntington's disease (HD) is caused by a CAG repeat trinucleotide expansion within the first exon of the huntingtin gene and causes a range of symptoms including motor, cognitive and psychiatric disturbances, which significantly affect daily activities, independence and quality of life, even during the early stages of the disease. Cognitive dysfunctions from early on in the HD disease process have been well documented and can include specific problems with attention, cognitive flexibility and memory. Indeed, difficulty sharing attention between more than one task has been demonstrated to be a specific and core deficit in HD.

   Cognitive training interventions, which focus on executive function, present a potentially exciting non-pharmacological treatment option for neurodegenerative diseases including HD. Studies in HD mice have previously demonstrated executive function impairments, including deficits in attention and subsequent studies have shown that cognitive training can benefit HD mice and prevent the onset of cognitive and motor disease symptoms. This work suggests that an early cognitive training intervention can have significant and long-lasting beneficial effects on HD symptoms. Although further systematic studies in mouse models of HD are required to inform the translational aspects of cognitive training interventions, these results provide important proof of principle evidence that cognitive training can provide benefit in mouse models of HD.

   Studies in human populations suggest that cognitive training, via repeatedly conducting tasks that require specific aspects of executive function such as attention, reasoning and memory, can improve cognitive function as people age. Computerised cognitive training studies have also been conducted in a number of neurodegenerative diseases including Parkinson's disease (PD) and Alzheimer's disease (AD). These studies have found that computerised cognitive training that can improve cognition in PD and AD. However, a systematic literature review of Europe PubMed Central using the keywords, 'Huntington's disease' and 'cognitive training' or 'cognitive therapy' or 'brain training' or 'executive function training' conducted from the years 1950 to 2015, produced 2 results. A review on cognitive burden in HD and a paper on exercise in a mouse model of HD benefiting cognitive symptoms. Thus, the use of cognitive training in HD is a considerably under researched area and to our knowledge cognitive training is yet to be explored in HD. Therefore, feasibility studies, such as the one proposed in this application are crucial in trialing novel potential therapeutic interventions.

   The outcome measures used to determine patient benefit in cognitive training studies can vary significantly between studies. Furthermore, this is the first time that such an intervention has been used in people with HD. Therefore, the outcome measures used in cognitive training studies to determine patient benefit need to be carefully explored and defined prior to beginning the study. The candidate outcome measures for use in this study have been chosen to include both cognitive and motor measures specific to people with HD to best evaluate the outcome of the intervention. Difficulty sharing attention has been shown to be a specific problem in HD. Attentional sharing can be measured clinically using dual tasks where participants are required to do two tasks at the same time. The two tasks can be from the same modality such as walking and carrying a tray, or from different modalities such as walking combined with a cognitive component such as counting. Dual task studies have shown that people with HD have reduced attentional sharing capacity, particularly when the dual task has a cognitive element. As the ability to complete dual tasks and increasing attentional demand are key skills in everyday life, deficits in such tasks can severely affect independence, increase the risk of falls and reduce quality of life. The proposed study will use dual task performance to assess feasibility, acceptability and to gather preliminary efficacy data on the effect of cognitive training interventions in people with HD.

   Environmental enrichment has been shown to improve disease symptoms in HD mice and a retrospective study regarding lifestyle of people with HD suggests that a passive or sedentary lifestyle, lacking in enriching activities, may contribute to earlier onset of disease symptoms. There is also preliminary evidence that motor training can produce functional benefits in HD and accumulating evidence of feasibility and functional improvements from both in- and out-patient exercise and rehabilitation programmes. Motor training exercise studies have shown that multi-modal exercise interventions are well tolerated and associated with improvements in movement, cognition and mood alongside increases in health related quality of life. Work is now ongoing to develop methods to support and enhance adherence to home exercise in HD. Furthermore, the investigators now have preliminary evidence that an intervention with both motor and cognitive components (a training regimen in which patients' train to drum increasingly complex rhythms to music) can produce improvements on the symbol digit modalities, a test of executive function, with accompanying changes on MRI tractography. Brain imaging studies are hugely important in greater understanding the biological mechanisms which may underpin any intervention in a neurodegenerative disease.

   Strategies for conducting cognitive training can vary between research studies. Some use taught exercises or puzzles which participants learn and then repeat. However, the utilisation of computerised cognitive training strategies provides several advantages over repeating practical tasks. Computerised cognitive training strategies are automated and can be completed by participants at their convenience, they provide automated tasks which require comparatively little movement to complete and provide several objective outcome measures. Furthermore, the specific HAPPYneuron cognitive training software that the investigators are using in this study provides an interface for the researcher to observe the progress of study participants and it can be made available in different languages to allow for consistent training globally. However, as this is a feasibility study, the computerised cognitive training intervention will be optimised taking into account the feedback and views of people with HD.
2. Study Aims The primary aim of this study is to determine if computerised cognitive training, is feasible and acceptable for people with HD. The researchers will investigate the familiarity of participants with the computerised cognitive training programme, its usability and determine key outcome measures for use in cognitive training studies, before conducting a randomised feasibility study. The randomised feasibility study will also explore the biological underpinnings of any observed behavioral changes using MRI scanning, this is an optional component of the study. During this study, important parameters will be established, which will allow us to develop the intervention programme for use in a larger patient cohort.

   2.1. Specific Objectives

   The objectives of the proposed study are to:

   (i) investigate the familiarity of participants ad usability of computerised cognitive training programmes and determine key outcome measures for use in cognitive training studies.

   (ii) assess the feasibility of delivering a home based computerised cognitive training programme for people with HD, considering:
   * The willingness of eligible participants to receive the intervention and participate in a feasibility study (including the feasibility of randomisation)
   * Potential barriers to recruitment or completion of the study
   * Response rates and adherence to the cognitive training programme (iii) determine any behavioural changes which may occur during the intervention or comparable control arm.

   (iv) use brain imaging techniques to explore the biological underpinnings of any observed behavioral change (optional).

   (v) evaluate the intervention using participant and family member/carer feedback to future use in this patient population.
3. Study Design Participants will be recruited from the Cardiff Huntington's disease Centre. Participants will be asked to complete a range of computer and paper based cognitive tasks, motor tasks and interviews in their first research visit, which may coincide with their ENROLL-HD visit. Participants will then be invited back to complete baseline assessments for the feasibility study within the next 4 weeks. After randomisation, those allocated to the intervention group will receive the 12-week home-based cognitive training intervention, supported by home visits and email or telephone reminders, as preferred. Those allocated to the control group will be asked to continue as normal although they will also receive home visits. At 6 weeks an optional MRI scan will be conducted in addition to cognitive tasks. 12 weeks after completing baseline assessments, participants will be invited back to complete the final outcome assessments.
4. Participant Selection The Cardiff HD Centre is an Enroll-HD (previously Registry) site and many patients attending the clinic are enrolled in this study (REC no. 04/WSE05/89). Patients already enrolled to a global Enroll-HD observational study will be invited to take part in this study. The progression of symptoms in these Enroll-HD participants are monitored longitudinally. One of the optional components within the Enroll-HD study is the giving of permission by participants to be contacted about other additional and affiliated HD research studies, and for their coded data to be accessed by researchers conducting HD related research. As such, a full clinical data set including full medical and medication history will be available for each research participant and this data may be used during the study. In addition, the investigators would like to gather the views of family members, friends and carers. Participants will be asked to provide consent so that the investigators can talk to their family member, friend or carer, who may be attending research visits with the participant, about their involvement in the study. If informed consent is obtained, via a participant dated consent form, the family member, friend or carer will be invited to be interviewed about the study.
5. Recruitment 5.1. Number of Participants This is an initial proof of principle study; thus no formal sample size calculations have been completed. The investigators will aim to recruit 50 participants with a target of randomising 40 participants. The suggested numbers are based on previous literature regarding cognitive training in other diseases and considering that MRI is an optional component of the study. The study team have funds for the MRI scanning of 16 participants during the study, scanning will be conducted on a first come first served basis and once the funds for scanning are used no further participants will be able to be scanned. This study is an essential step towards a larger systematic study of cognitive training and will inform the design and delivery of such a trial, as well as providing data to inform a power calculation to estimate sample size in the future.

   5.2. Recruitment Process Potential participants, who have already consented to participate in ENROLL-HD may be approached during their clinical visits and will be informed of the study. Potential participants will receive an information sheet about this study and be will be given sufficient time to ask questions and discuss the study with the researcher. If required, potential participants can take the information sheets home and discuss the study with their family and friends. Potential participants who wish to consent will be reminded that they can change their mind or withdraw without reason at any time. If the potential participant is willing to proceed with the study, they will be asked to sign a consent form and the study assessments will begin.

   5.3. Informed Consent The participant will be allowed as much time as needed to consider the Participant Information Sheet (PIS) and the opportunity to question the research team or independent parties to decide whether he/she will participate in the study. All participants will have the procedures explained in detail, including that the study design is randomised, that MRI scanning is an optional component and that they can withdraw at any time. Informed consent will then be obtained by means of participant dated signature and dated signature of the person who presented and obtained the informed consent. The original signed form will be retained at the study site. After informed consent has been received the first study visit will take place. Participants will be reminded that they can withdraw from the study at any time, without the need to give a reason and this will not affect their current or future care. Participants will be asked during the consent process if their family member or carer can be asked their opinions of cognitive training interventions, this is an optional component of the consent form. If consent is provided to ask family members, friends or carers that attend the clinic with the participant, they will be asked to read a separate information sheet. If they agree to participate, they will be asked to sign a consent form and they will then be interviewed regarding the study.

   5.4. Health Checks/Screening Required for Magnetic Resonance Imaging (MRI) Scanning MRI scanning is an optional component of the study. Thus, as part of the pre-screening process, all participants will be screened for contraindications to MRI. In addition, comprehensive screening for MRI contraindications will be completed immediately before each MRI scan by the researcher and the MRI operator before the participant is allowed into the scanning room.

   5.5. Randomisation Procedures As the study includes an intervention and control group, randomisation will be performed using a minimisation procedure and programme to ensure balance between the groups for categorical variables of age and cognitive function. Minimisation will be performed by the researcher, considering age and cognitive results of the most recently published global ENROLL-HD study data. Age and cognitive function will be given the same weighting during the minimisation procedure. Age will be classified into two categories: 1) < 45 years and 2) > 45 years. The total cognitive score of the participant in the Categorical Verbal Fluency Test, will be used to classify participants into two categories. The randomisation procedure will be carefully explained to all potential research participants and is specifically outlined in both the PIS and CF. Randomisation will only be performed after the participant has signed the CF and completed the initial and baseline assessments. Participants allocated to the control group will be asked to carry on as normal. Once allocated to a group, participants will receive an allocation letter detailing the group that they have been randomised to. Unfortunately, due to licencing restrictions those allocated to the control group will only be able to use the cognitive training software in the first research visit and during the baseline and outcome assessments of the second and third research visits. It will be made clear to all potential participants at the end of the study, they will have to stop using the cognitive training software as their access to the login system will expire.
6. Study Procedures

   6.1 The 12-week Cognitive Training Intervention The 12-week cognitive training intervention will be completed in participant homes. The intervention will be supported by email, text and telephone reminders (as preferred by the participant and detailed in the Case Report Form) and home visits. Home visits will be conducted for both the active and control groups. Although additional home visits may be necessary if a participant is concerned about using the software. During the research visits, for the active group, the researcher will ensure that the participant is comfortable with the software, offering support and guidance and a battery of cognitive assessments will be performed. For the control group during home visits the researcher will complete the cognitive test battery and talk to the participant about their day. The intervention is designed to be conducted with minimal supervision and this is something that will be explored during participant and friend, family member or carer interviews. When completing home visits, the researcher will comply with the Lone Workers Policy in existence at the Cardiff HD Centre and will discuss visits with the research team prior to completing them to ensure that safety is not compromised at any time. Participants will be asked to complete the training programme provided using HAPPYneuron software for a minimum of 30 minutes 3 times a week for 12 weeks. After the participant completes the 30 minute training programme they will be free to complete any other of the 'games' available on the HAPPYneuron computerised cognitive training software. Completion of the cognitive training programme will be monitored and supported using email or telephone reminders (as preferred by the participant) and home visits by the researcher. This will allow patient adherence with the cognitive intervention programme to be monitored and therefore the feasibility and acceptability of the programme by the participant to be explored. Each participant will be provided with a unique log in. The software provides an interface that allows the researcher to track the regularity of use and progress of all study participants. Therefore, the investigators will be able to remotely determine how often and for how long participants are using the software and can analyse participant performance on each cognitive task. Furthermore, the performance of participants for each specific task, during each cognitive training session is measured and can be used to determine improvements in specific cognitive tasks, for example in response accuracy or response time, throughout the study. Participants will be made aware that the researcher is able to see their training activity throughout the study.

   The cognitive training software the investigators plan to use in this study is easy to use, is automated, provides non-biased data recording, provides an interface which allows the researcher to track compliance remotely. It has previously been validated in both healthy controls and patients with depression, and has shown patient benefit including improved cognition and functionality. At the end of the study the participant login details will expire and they will no longer be able to access the cognitive training software, this is made clear in the PIS. The intervention is designed to be completed independently, although in this feasibility study, with the agreement of the participant, the investigators will be specifically exploring the involvement of any friends, family members of carers using semi-structured interviews at the beginning and end of the study.

   6.2. Magnetic Resonance Imaging (MRI) Scanning Cardiff University has a world leading brain imaging research centre (CUBRIC) which provides access to state of the art research facilities and equipment. Therefore, MRI scanning will be used in this study, as an optional component, to greater explore the biological effects if any, that the cognitive training programme may have. Prior to consent, potential participants will be screened for any contradictions to MRI. Further screening will be conducted prior to any MRI scanning procedures. MRI scanning is an optional component of the feasibility study, therefore if participants cannot or do not want to undergo the MRI scanning procedures, they will still be able to take part in the study. Participants will also be made aware that they are free to withdraw from the MRI scanning component of the study at any time, without the need to give a reason and this will not affect the care that they receive.

   If a participant consents to MRI, the MRI scanning procedure will be carefully explained and discussed with the participant and the participant will have the opportunity to experience the 'mock' MRI scanner, if they feel this may be helpful. The MRI scan will be conducted at a research visit 6 weeks into the intervention. An MRI scan will then be conducted by a fully trained MR Operator with the help of a researcher who is MR safety trained. The scan will be acquired on a 3T Siemens Prisma scanner with 32 head coils. The MRI scanning protocol will include scans to assess a structural scan to assess gross macrostructure, microstructural scans to assess white matter and myelination changes as well as quantitative fMRI to measure resting cerebral blood flow. The complete scanning protocol is expected to last no longer than 90 minutes, but will be led by the participant to ensure that they are comfortable throughout the scanning procedure.
7. Data Collection For the majority of assessment procedures, data will be collected on paper data collection forms and the results of the tests subsequently transferred to a secure online database. The data in the online database will be verified against the paper form to ensure data integrity. Original data collection sheets will be filed and stored securely in the TMF.

   For the semi-structured interviews, questions will be asked orally by the researcher, audio recorded and transcribed verbatim. Although some flexibility may be necessary to avoid the need for protocol amendments. A list of topics to be included in the interview schedule for participants and family members, friends or carers who attend the research visit with the participant include:
   * How the intervention is perceived/was received?
   * Expected or perceived impact on daily routine
   * Expected or perceived impact on family members/ carers
   * Overall expectations
   * Expected or perceived acceptability (support or help required)
   * Thoughts and views on the randomisation procedure
   * Potential barriers to completing the intervention
   * General views or comments on the cognitive training intervention
8. Data Analysis As the proposed study is a feasibility study for the use of computerised cognitive training for people with HD, the study is not formally powered. The primary aim is that of feasibility, so eligibility, recruitment and acceptability of the study will all be evaluated. Adherence to the proposed cognitive training intervention and any adverse effects will also be reported. Therefore, crucial inferences will be made which will allow an estimation of parameters that can inform definitive and future trials in this specific patient population.

   8.1. Statistical Analyses Summary statistics of demographics (age, gender, height and weight) and disease burden scores will be reported. Descriptive data will include an evaluation of eligibility, recruitment, retention rates and acceptability of, and adherence to the intervention, with 95% confidence intervals. The completion of outcome measures and assessments will also be reported. Graphical illustration will be used to check distributions of outcome data.

   Successful adherence to the intervention will be defined as having completed 12 weeks of the computerised cognitive training for a minimum of 3, 30 minute sessions per week. This is a feasibility study; thus an estimation of retention rates may be difficult with such as small sample size. Therefore, it is suggested that if retention rates are greater than 75%, the investigators will consider this intervention to be feasible. If the proportion retained is less than this but greater than 65%, the investigators will consider adjusting the intervention to increase this in future investigations. The qualitative work will help to establish why retention rates are as they are at the end of the study. A retention rate lower than this would require substantial changes to the intervention and therefore would require further piloting and feasibility studies. Changes in the outcome assessments in will be analyzed using analysis of covariance (ANCOVA) with the baseline score of that variable in addition to the balancing variables (age and UHDRS TMS) as covariates.

   Data collection will be performed via HAPPYneuron software systems and initially on data collection forms before transfer to a database. Data completeness will be monitored at the point of collection; therefore, the investigators do not expect large amounts of missing data. As it is our intention to inform future confirmatory trials, the investigators will explore the feasibility of outcomes as applied in this trial and this population. The investigators will consider internal reliability of all outcome measures, as some have not been previously used in HD or applied to computerised cognitive training interventions.
9. Dissemination The research team are committed to disseminating the research findings to the general public and patient groups and will seek to present the results at patient open days, engagement events and outreach activities. Dissemination is a particular passion of the CI. Furthermore, in order to communicate the research widely, the results may be disseminated via social media, through newsletters and other patient engagement outlets in appropriate language and format for the general public to understand. If a participant indicates that they would like to be informed of the results of the trial a report of the findings will be sent to them at trial closure. Where results are presented, they will always be presented in such a way that data from individual participants cannot be identified. In addition to the significant public and patient outreach dissemination, the research findings will be written up for publication in a scientific journal. The results may also be presented at scientific meetings, or in talks at academic institutions.
10. Data Storage, Handling, Retention and Confidentiality All data will be stored within a firewall and password-protected computer system within a swipe-card secured building. Researchers associated with the study will have confidential access to files, which allow the matching of recorded data to participants. No data, whether paper or electronic, will leave Cardiff University sites without being completely anonymised, i.e., all identifiable data will be removed from the dataset. Any electronic files or disks will be stored on Cardiff University sites and electronically on Cardiff University systems. At the conclusion of the study identifiable data will be destroyed and non-identifiable data will be archived, although it will still be accessible to the study team. Data will be archived for 15 years, in line with Cardiff University policies and procedures. Study data may be shared with the organisation funding the study. Where data leaves Cardiff University it will be strictly anonymised. Anonymised data may be shared with researchers at other organisations in the UK or overseas and it may be made publicly available for future research use. In the case of the data generated using HAPPYneuron systems, this data is captured centrally and stored outside of the Cardiff University systems and is therefore subject to HAPPYneuron's policies and procedures. However, a subset of this data will be extracted for use in the study and transferred on to Cardiff University systems as described above.

    All participant identification and referral procedures as well as procedures for data storage, processing and management will comply with the Data Protection Act 1998. Data will be kept for 15 years in line with Cardiff University's Research Governance Framework Regulations for clinical research. This data will be stored confidentially on password protected servers maintained on the Cardiff University Network. Data will be stored in locked cabinets and/or on secured computer hard-drives (password protected) in an access controlled building and will be retained indefinitely. This is in compliance with the guidelines set by the Cardiff University Research Governance Framework. The confidentiality of participants will be preserved in accordance with the Data Protection Act 1998. All participants will be allocated an Enroll-HD unique study number identifier and in the case of family members, friends or carers, they will be allocated a unique study number in relation to the participant. All data collected will be held in a linked anonymised form.
11. Study Closure Definition The end of study is the date of the last visit of the last research participant.
12. Indemnity Cardiff University will provide indemnity and compensation in the event of a claim by, or on behalf of participants, for negligent harm as a result of the study design and/or in respect of the protocol authors/research team. Cardiff University does not provide compensation for non-negligent harm.
13. Sponsorship Cardiff University will act as sponsor for this study.
14. Funding

The study is funded by two research grants:

1. 18 month research grant from the Jacque and Gloria Gossweiler Foundation, awarded to Dr. Emma Yhnell (Lead Applicant), Prof. Anne Rosser, Prof. Monica Busse and Dr. Claudia Metzler-Baddeley. 'Exploring cognitive training as a non-pharmaceutical therapeutic intervention for people with Huntington's disease.' (funding start date: 1st April 2016, study end date: 30th September 2017).
2. 36 month fellowship award to Dr. Emma Yhnell from Health and Care Research Wales. 'Using computer based cognitive training to provide a personalised therapeutic intervention for people with Huntington's disease.' (funding start date: 1st October 2016, study end date: 30th September 2019).

15. Study Management The project will be managed by the CI Dr. Emma Yhnell, with the support of colleagues from the Cardiff HD Centre, including Ms. Hannah Furby, Prof. Monica Busse (SEWTU), Prof. Anne Rosser (Clinical Responsible for Care) and Dr. Claudia Metzler-Baddeley (CUBRIC). In addition the CI will receive advisory support from members of SEWTU, in the form of monthly research meetings and email support for the duration of the project. The SEWTU advisory board includes: Dr Rachel Breen, Dr. Rebecca Playle, Mr. Gareth Watson and Dr. Lucy Brookes-Howells.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HD diagnosis by genetic test.
* Over 18 years of age.
* Enrolled in the EHDN Registry/Enroll-HD study.
* Stable medication regime 4 weeks prior to recruitment (and not anticipated to change medications during the study period).

Exclusion Criteria:

* Inability to provide consent.
* Any known neurological condition (other than HD).
* Currently actively involved in any other interventional trial (i.e. have begun the intervention) or within four weeks of completing the final assessments of an interventional trial.
* Currently regularly completing computerised brain training programme.
* MRI contraindications (e.g. a pacemaker) as established using standard screening procedures (optional).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2019-03-13 (Actual); Study Completion 2019-03-13 (Actual)

PRIMARY OUTCOMES:
Number of participants able to complete the feasibility study as measured by retention rate | During 3 year study (Outcome Measure)
  The primary outcome measure of this study is feasibility for this patient group, a retention rate of 75% will be considered feasible.

SECONDARY OUTCOMES:
Number of participants able to complete computerised HAPPYneuron pro cognitive training as assessed by task performance and the quality of the data generated. | During 3 year study (Outcome Measure)
  The cognitive training programmes completed will be assessed. The level of achievement and quality of the data generated will be assessed.
Symbol digit modality test | During 3 year study (Baseline Assessment and Outcome Assessment)
  This is a simple substitution task to measure executive functioning. Using a reference key, the participant has 90 seconds to pair specific numbers with given geometric figures.
Stroop tasks on paper of colour and work naming | During 3 year study (Baseline Assessment and Outcome Assessment)
  In the stroop tasks, the participant is required to read words of colour names (e.g. red, blue) printed in black ink, and is asked to identify colours. This trial is intended to rule out colour blindness and ensure an adequate reading ability to complete the task. In the second stroop baseline trial, the subject must name the colour in which a word is presented, while ignoring the printed word. Thus, incongruence between the words colour and identity requires inhibition and response selection.
Categorical verbal fluency (letter and categorical fluency test) | During 3 year study (Baseline Assessment and Outcome Assessment)
  The fluency tasks require participants to verbally generate words beginning with a given letter (e.g. words beginning with the letter F) or category (e.g. animals). Participants are given one minute to retrieve as many words as possible and are instructed to avoid repetitions.
Trail making A and B tests | During 3 year study (Baseline Assessment and Outcome Assessment)
  This pencil and paper task uses randomly placed letters (and numbers for part B) as stimuli and participants must connect in sequence by drawing a continuous line with a pencil (e.g. from A-1-B-2-C-3 for part B). There is a brief sample for instruction purposes.
Digit Span Forward subtest from Weschler's Adult Intelligence Scale (WAIS) | During 3 year study (Baseline Assessment, During Intervention and Outcome Assessment)
  This task of working memory involves the participant being read a sequence of numbers and is asked to recall the numbers in the same order.
Dual-tasking. Subjects are required to switch their attention between two competing tasks. Subjects will be asked to cross out a series of boxes whilst simultaneously recalling a digit sequence. | During 3 year study (Baseline Assessment, During Intervention and Outcome Assessment)
  This test requires subjects to switch their attention between two competing tasks. Subjects will be asked to cross out a series of boxes whilst simultaneously recalling a digit sequence at a difficulty matched to their own digit span length.
Tower of Hanoi | During 3 year study (Baseline Assessment, During Intervention and Outcome Assessment)
  The Tower of Hanoi task has been used extensively as a test of planning ability in neuropsychological patients and normal populations to assess executive function. Participants are asked to preplan mentally a sequence of moves to match a start set of discs to a goal, and then to execute the moves one by one.
Card sorting task of executive function | During 3 year study (Baseline Assessment, During Intervention and Outcome Assessment)
  This is a neuropsychological test of "set-shifting", i.e. an executive function that reflects mental flexibility in the face of changing schedules of reinforcement. It requires subjects to identify a rule (e.g. a commonality between cards) and sort cards into groups according to that rule.
Number of participants able to fully complete timed up and go (TUG) motor assessments as assessed by time taken to complete the task | During 3 year study (Baseline Assessment, During Intervention and Outcome Assessment)
  The Timed Up and Go Task (TUG) will be used to determine participant mobility and balance. The task will involve the participant rising from a seated position, walking 3 metres and returning to a seated position. A quantitative version of the task and a dual task will also be performed.
Participant scores in the 'money box test' | During 3 year study (Baseline Assessment and Outcome Assessment)
  The money box test has been developed as a dual task for use in HD to assess upper limb dexterity and motor function.
MRI scanning results | During 3 year study (Baseline Assessment, During Intervention and Outcome Assessment)
  The MRI scanning protocol will include scans to assess a structural scan to assess gross macrostructure, microstructural scans to assess white matter and myelination changes as well as quantitative fMRI to measure resting cerebral blood flow.
Participant scores on the Hospital Anxiety and Depression Scale (HADS) | During 3 year study (Baseline Assessment, During Intervention and Outcome Assessment)
  This short scale will be used to screen for depression and anxiety symptoms.
Participant scores on The International Physical Activity Questionnaire (IPAQ) | During 3 year study (Baseline Assessment, During Intervention and Outcome Assessment)
  This questionnaire assesses physical activity undertaken across a comprehensive set of domains including leisure time, domestic and gardening activities, work-related and transport-related activity.
Participant scores on HD-Pro-TriadTM Questionnaire | During 3 year study (Baseline Assessment, During Intervention and Outcome Assessment)
  This is a reliable and valid health-related quality of life instrument that captures the typical triad of HD symptoms.
Participant scores on the Life-Space Assessment | During 3 year study (Baseline Assessment, During Intervention and Outcome Assessment)
  This tool can be used to establish the spatial extent of a person's mobility a useful outcome measure of independence.

OTHER OUTCOMES:
Qualitative experiences of participants and nominated carers, friends or family members. | During 3 year study (Baseline Assessment and Outcome Assessment)
  Analysis will provide key words which will elicit general themes and attitudes to the cognitive training intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiff University, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be made available.

REFERENCES:
- [Derived] Yhnell E, Furby H, Lowe RS, Brookes-Howell LC, Drew CJG, Playle R, Watson G, Metzler-Baddeley C, Rosser AE, Busse ME. A randomised feasibility study of computerised cognitive training as a therapeutic intervention for people with Huntington's disease (CogTrainHD). Pilot Feasibility Stud. 2020 Jun 19;6:88. doi: 10.1186/s40814-020-00623-z. eCollection 2020. PMID 32577299
- [Derived] Yhnell E, Furby H, Breen RS, Brookes-Howell LC, Drew CJG, Playle R, Watson G, Metzler-Baddeley C, Rosser AE, Busse ME. Exploring computerised cognitive training as a therapeutic intervention for people with Huntington's disease (CogTrainHD): protocol for a randomised feasibility study. Pilot Feasibility Stud. 2018 Feb 6;4:45. doi: 10.1186/s40814-018-0237-0. eCollection 2018. PMID 29445514